CLINICAL TRIAL: NCT01734577
Title: The Effect of Trigger Point Dry Needling to the Multifidus Muscle on Resting and Contracted Thickness of Transversus Abdominis in Healthy Subjects
Brief Title: Effect of Dry Needling Multifidus on Thickness of Transversus Abdominis in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Emilio, Dr. Emilio J. Puentedura, University of Nevada, Las Vegas
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: UNLVPT-4059
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Back Pain
Keywords: Back pain
MeSH Terms: conditions — Back Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dry needling (Active Comparator): Monofilament needles will be inserted into each subject's left multifidus muscle and stimulated mechanically for a local twitch response
  Interventions: Procedure: Dry needling
- Sham needling (Sham Comparator): Monofilament tubes will be pressed into the left multifidus muscle and mechanically manipulated to give the sensation that needling is occuring.
  Interventions: Procedure: Sham needling

INTERVENTIONS:
Procedure: Dry needling — Sterile monofilament needles
  Arms: Dry needling
Procedure: Sham needling — Applicator tubes from the sterile monofilament needles
  Arms: Sham needling

SUMMARY:
Intramuscular therapy (also known as dry needling) has been shown to give dramatic relief of musculoskeletal pain. The mechanisms of action remain unknown, and this study will examine for a neurophysiological effect.

DETAILED DESCRIPTION:
Consenting adults will be taught how to contract their abdominal muscles, and to contract transversus abdominis in particular. They will then have real time ultrasound measurements of the resting and contracted thickness of their left transversus abdominis muscle. After this, they will receive actual or sham needling to their left multifidus muscle by another researchers blinded to the real time ultrasound measurements. After needling or sham intervention is complete, the original researchers will return to re-measure transversus abdominis. They will be blind to intervention allocation.

ELIGIBILITY:
Inclusion Criteria:

* Age, absence of back pain or symptoms for greater than 6 months and ability to perform DCC. Subjects must also report they are comfortable with being 'needled'.

Exclusion Criteria:

* Presence of back pain or symptoms within the last 6 months, history of: abdominal or spinal surgery, significant scoliosis, rheumatoid arthritis, osteoporosis, osteopenia, active ankylosing spondylitis. If a subject reports a fear of needles.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Thickness of transversus abdominis at rest and during contraction | 1 day
  Real time ultrasound measurement

CONTACTS AND LOCATIONS:
Overall Officials: Daniella Morton, BSc, Study Director — University of Nevada Las Vegas Physical Therapy; Sarah Buckingham, BSc, Study Director — University of Nevada Las Vegas Physical Therapy; Crystal Montoya, BSc, Study Director — Univesity of Nevada Las Vegas Physical Therapy
Locations (1):
- University of Nevada Las Vegas - Department of Physical Therapy, Las Vegas, Nevada, United States

REFERENCES:
- [Derived] Puentedura EJ, Buckingham SJ, Morton D, Montoya C, Fernandez de Las Penas C. Immediate Changes in Resting and Contracted Thickness of Transversus Abdominis After Dry Needling of Lumbar Multifidus in Healthy Participants: A Randomized Controlled Crossover Trial. J Manipulative Physiol Ther. 2017 Oct;40(8):615-623. doi: 10.1016/j.jmpt.2017.06.013. PMID 29187313